CLINICAL TRIAL: NCT04802135
Title: Creation of a Register of Patients With Neonatal-onset Epileptic Encephalopathy
Acronym: IMPROVE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-51; ID-RCB (Other: 2020-A01363-36)
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Epileptic Encephalopathy
Keywords: EOEE; epilepsy; KCNQ2
MeSH Terms: conditions — Epilepsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — directive questionnaire administered during an individual face-to-face interview

SUMMARY:
Electrical activity emerges in the third trimester of pregnancy, plays an important role in the construction of cortical maps, and is impaired in patients with severe early epileptic encephalopathies (EOEE). EOEE are rare and severe epileptic syndromes characterized by epilepsy that begins within the first three months of life and is associated with rapid deterioration of motor, cognitive and behavioral skills.

There is a genetic basis for the EOEE. Together with other laboratories, the investigators have identified de novo pathogenic variants in the KCNQ2 gene encoding the Kv7.2 subunit of the Kv7 / M potassium channel, a channel known to control neuronal excitability in the brain and spinal cord. via the current M (IM). Pathogenic variants of the KCNQ2 gene represent the main cause of EOEE and the term KCNQ2-related epileptic encephalopathy (KCNQ2-REE) is now used to define this condition.

KCNQ2-REE patients have a remarkably homogeneous phenotype at the start, with epilepsy that begins in the first days after birth, seizures that result in tonic muscle spasms that last from 1 to 10 seconds, and an interictal EEG called "suppression-burst". "That is, paroxysmal bursts of activity interspersed with periods of electrical silence. In this group, more than 50% of the patients present a remission of the epilepsy and a quasi-normalization of the EEG which can occur a few weeks to several months after the onset of the seizures. Despite this positive evolution in terms of seizures, the developmental progression is abnormal and the phenotype is severe with an absence of language, autistic behavior and a subsequent development of motor disorders such as diplegia, spasticity, ataxia or dystonia.

The ambition of this project is to increase knowledge of epileptic encephalopathies linked to KCNQ2 at the clinical and molecular levels, to decipher the pathophysiological mechanisms and to propose therapeutic strategies.

This project aims to better describe the clinical, EEG, imaging, developmental and long-term follow-up characteristics of patients carrying the KCNQ2 mutation identified in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy beginning before 1 month of life, and requiring the initiation of anti-epileptic treatment
* Without occasional cause
* Without brain malformation explaining epilepsy
* No opposition from parents / guardians
* Possibility for parents to complete parent questionnaires

Exclusion Criteria:

* Neonatal attacks of occasional cause (glycemic disorder, infection, etc.)
* Acquired neonatal epilepsy (post-anoxic encephalopathy, stroke sequelae, etc.)
* Neonatal epilepsy related to a brain malformation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective observational study initially then prospective with inclusion of all patients with a KCNQ2-REE whose diagnosis was made in the EPIGENE network
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-06 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
importance of the developmental disorder | Month 36
  Developmental quotient
definition of the active phase of epilepsy | Month 36
  Presence of at least monthly seizures and interictal EEG showing paroxysmal abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier Arnaud, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (15):
- France (15):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - Hospices Civils Lyon, Lyon
  - Hôpital La Timone, Marseille
  - CHU Montpellier, Montpellier
  - APHP Pitié Salpêtrière, Paris
  - APHP Robert Debré, Paris
  - Hôpital Necker, Paris
  - CHU Rennes, Rennes
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No